CLINICAL TRIAL: NCT05670340
Title: Effect of Bone-related and Soft-tissue-related Variables on the Marginal Bone Loss of Platform-matched and Platform Switched Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Full Professor in Prosthodontics, University of Salamanca
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Usal_2020_433
Record Dates: First submitted 2022-11-29; First posted 2023-01-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dental Implant; Soft Tissue; Partial-edentulism; Bone Loss
Keywords: dental implant; marginal bone loss; peri-implant soft tissue; ISQ
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: The implant abutment height could be short (<2mm) or long (>2mm)
Who Masked: Participant, Outcomes Assessor
Masking Description: only the care provider knows the group asignement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swithed-platform (Experimental): In this group the implants will be rehabilitated with a narrower emergence profile for the prosthetic rehabilitation.
  Interventions: Device: Switched Prosthetic Profile
- Matched-platform (Active Comparator): This the conventional approach in wich the prosthetic rehabilitation is matched with the implant-platform dimensions
  Interventions: Device: Matched Prosthetic Profile

INTERVENTIONS:
Device: Switched Prosthetic Profile — The implant will be rehabilitated with a switched emergence profile
  Arms: Swithed-platform
Device: Matched Prosthetic Profile — The implant will be rehabilitated with a matched emergence profile
  Arms: Matched-platform

SUMMARY:
In this clinical trial the effect of the implant-abutment morphology (platform-switched vs platform matched) will be assessed in both soft tissue (soft tissue thickness) and hard tissue (marginal bone loss) outcomes. Several clinical predictors (initial implant position level, gingival biotype, abutment height and prosthetic emergence profile) will also be taken into account as modulating factors of the clinical outcome.

DETAILED DESCRIPTION:
This prospective clinical trial is conducted at the Dental Clinic of the Faculty of Medicine of the University of Salamanca. The protocol was developed in accordance with the 1975 Declaration of Helsinki, and later approved by the Bioethics Committee of the University of Salamanca with the number (Ref:473/2020)

Before initiating any procedure, each patient received information about the study design and signed an informed consent. The subjects are recruited consecutively following the admission protocols of the Dental Clinic of the Faculty of Medicine of the University of Salamanca, Salamanca, Spain. The inclusion criteria are:

(1) Patients of legal age (>18 years); (2) in need of at least one maxillary or mandibular dental implant to be inserted in mature bone (more than 4 months after tooth extraction) in the posterior area (premolars and molars); (3) with good oral hygiene (plaque and gingival index ≤ 25%). The exclusion criteria included clinical conditions that contraindicated implant surgery, (1) patients with immunological alterations, pregnant and lactating, (2) heavy smokers > 20 cigarettes/day, (3) with the need for bone or soft tissue augmentations, (4) patients whose anatomy prevented the correct three-dimensional placement of the implant to perform prosthetically guided screwed restorations.

All implants were placed by an experienced implantologist following standard procedures and the manufacturer's recommendations. All implants were connected to a transmucosal abutment to heal in one-stage approach. Several variables were collected in this surgical phase (bone quality, implant stability, implant-bone level, mucosal thickness, keratinized mucosa width ...)

After 3 to 4 months of implant healing all the clinical parameters were reevaluated and the final impression will be used for the manufacturing of a porcelain-fused to metal screwed crowns.

Two types of data will be analyzed: Cross-sectional and longitudinal data. On the one hand, cross-sectional data included sociodemographic (sex and age), behavioral (smoking, oral hygiene..) clinical (antagonist, adjacent dentition, arch location, implant diameter and length, insertion torque values, bone density, implant-level...) and prosthetics (abutment and prosthetic profiles, interocclusal prosthetic space, cantilever lengths...).

On the other hand, the longitudinal variables were classified into 2 types, related to the gingival tissues and related to the surrounding bone. Regarding the gingival tissues these were the longitudinal variables assessed in different follow-up observations (at 3, 6 and 12 months): plaque and gingival index, keratinized mucosa width. Regarding the bone-related variables the implant stability by ISQ as well as the marginal bone position were also measured at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (>18 years).
* With rehabilitation needs with 1 maxillary or mandibular implant in mature bone (more than 4 months after tooth extraction) in the posterior sector (premolars and molars).
* With good hygiene (plaque and gingival index ≤ 25%).

Exclusion Criteria:

* Medical conditions that contraindicated implant surgery.
* Patients with immunological alterations, pregnant and lactating.
* Heavy smokers > 20 cigarettes/day,
* Requiring bone augmentations or of soft tissues.
* Patients whose anatomy prevented the correct three-dimensional placement of the implant to perform prosthetically guided screw-retained restorations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the Peri-implant Marginal Bone level | At baseline (reference), in comparison with 3, 6 and 12 months
  The implant-bone level is assesssed radiographicly
Change in the Implant stablity quotient | At baseline (reference), and in comparison with the 3 months follow-up
  The ISQ is assesssed by Osstell
Change in the Gingival Thickness | At baseline (reference) and in comparison with the 3, 6 and 12 months follow-up
  The gingival thickness will be assessed by measuring the keratinized region around implants with a periodontal probe and a thickness caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Javier Montero, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quispe-Lopez N, Guadilla Y, Gomez-Polo C, Lopez-Valverde N, Flores-Fraile J, Montero J. The influence of implant depth, abutment height and mucosal phenotype on peri-implant bone levels: A 2-year clinical trial. J Dent. 2024 Sep;148:105264. doi: 10.1016/j.jdent.2024.105264. Epub 2024 Jul 23. PMID 39053878